CLINICAL TRIAL: NCT05219955
Title: Caregiver Stress and Sleep Study
Acronym: CARES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Stephen Smagula, Assistant Professor of Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: STUDY21100123; MH125846 (Other Grant/Funding Number: National Institute of Mental Health (NIMH))
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Depressive Symptoms; Caregiver Burden
Keywords: Depression; Caregiving; Late-Life; Morningness
MeSH Terms: conditions — Depression; Caregiver Burden

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active condition (SAMM Protocol) (Experimental): The goal of the SAMM protocol is to increase morning activity engagement over a 6-week period. Participants in this condition will review their morning routine, and make a list of potential morning activities to add. They will choose one activity and develop a plan for doing it. Each day, participants are asked to track if they do the morning activity plan. If unsuccessful, at weekly follow-ups, participants are asked to refine their plan or make a new one.
  Interventions: Behavioral: Morning Action Plan Execution; Behavioral: Activity Strategy-based Session with Therapist; Behavioral: Advance sleep-wake time
- Attention-matched supportive control condition (Active Comparator): Participants in this condition will receive sessions in the same number and duration as the SAMM experimental condition. Therapists will create a comfortable environment by demonstrating interest, empathy, and acceptance without judgment. Caregivers will be encouraged to talk about stressors they experience, providing an opportunity to voice and self-address their problems. In this control condition, therapists will not deliver any particular strategy except for active listening and referring to the educational materials.
  Interventions: Behavioral: Attention-based Session with Therapist

INTERVENTIONS:
Behavioral: Morning Action Plan Execution — Each day, participants are asked to track if they do the morning activity plan.
  Arms: Active condition (SAMM Protocol)
Behavioral: Activity Strategy-based Session with Therapist — Participants will meet weekly with a trained therapist to discuss their prescribed activity plan. If unsuccessful, at weekly follow-ups, participants are asked to refine their plan or make a new one. Each session lasts about 30-45 minutes.
  Arms: Active condition (SAMM Protocol)
Behavioral: Attention-based Session with Therapist — Participants will meet weekly with trained a therapist to talk about stressors they experience, providing an opportunity to voice and self-address their problems. In this control condition, therapists will not deliver any particular strategy except for active listening and referring to the educational materials
  Arms: Attention-matched supportive control condition
Behavioral: Advance sleep-wake time — Some participants will be asked to adjust their sleep schedule to accommodate morning activity engagement by introducing or altering mechanisms known promote early rising (i.e., light exposure, reward and processes, etc.)
  Arms: Active condition (SAMM Protocol)

SUMMARY:
This study includes a randomized experimental component where therapists will systematically deliver an experimental behavioral probe or a supportive control condition. The aim is to evaluate effects on meaningful health-relevant measures including morning activation levels, depression symptoms, rumination, and aspects brain connectivity previously linked with depression.

DETAILED DESCRIPTION:
Depression symptoms are a major public health concern in family dementia caregivers (dCGs) with shared risk factors. With more people living with dementia in the coming decades, more people will become unpaid dCGs. Replacing dCGs with skilled workers is untenable and would cost an estimated $162 billion annually. An estimated 1 in 5 dCGs have a depressive disorders. Over periods of 1-2 years, studies estimate that 25-48% of dCGs will develop new clinically significant symptoms or disorders. Depression symptoms relate to poorer quality caregiving and have health implications, including increased risk for physical function decline and chronic disease mortality. Especially when other risk factors are present, depression symptoms increase the likelihood that symptoms will worsen and disorders emerge. As in older adults generally, the recent National Academies of Sciences, Engineering, and Medicine report "Families Caring for an Aging America" states that the impact of caregiving on mental health is "highly individual," i.e., allocated to caregivers with vulnerability factors. This study focuses on one such vulnerability, morning activation deficits (MADs), based on evidence that MADs are a promising modifiable target for precision depression interventions in dCGs.

Investigators recently observed that MADs predict the depression symptoms persistence, independent of other key factors in dCGs. Data from dCGs shows that the relationship between MADs and depression symptoms involves heightened resting-state amygdala-posterior cingulate connectivity. In the context of prior literature, this implicates rumination. Given that bi-directional relations are plausible, controlled experimental data are needed to determine if targeting morning inactivation influences depression's mechanisms. If so, this would confirm MADs as a clinically actionable intervention target for controlling associated depression mechanisms.

Investigators piloted targeting MADs by using activity scheduling and monitoring, the logically relevant component of existing approaches, which is called Scheduling Activity and Monitoring Mornings (SAMM). MADs are defined as difficulty "getting going" and related objective morning inactivity. The SAMM protocol aims to increase the ease/level morning activity engagement by making, scheduling, and monitoring a morning action plan. Pilot data demonstrates that SAMM engages the target (MADs) and affects mood. This support the feasibility of using SAMM to probe effects of target modification on the hypothesized (ruminative processes) and alternative pathways. Tracking effects of modifying MADs with multi-modal data will elucidate how MADs may contribute in depression's mechanism. This randomized controlled study is needed to determine if SAMM has causal effects apart from non-specific therapeutic effects. Results will indicate if/how targeting MADs with SAMM could be pursued in precision efficacy trials.

Investigators are not proposing a prevention or treatment efficacy trial. The overarching aim is to delineate a mechanism that investigators propose operates across continuums of depression severity, risk, and resilience. Aim 1 will compare dCGs selected to be on either end of a spectrum: dCGs with MADs at levels linked with depression symptoms versus "morning type" dCGs who habitually prefer morning activity engagement. This provides a window into the mechanism by which MADs predict depression symptom persistence, while being a "morning type" appears protective. This contrasts with the designs of depression risk/incidence, prevention efficacy, and treatment efficacy studies; such studies select participants based on depression thresholds, which here, would restrict natural variability in (and bias estimates of) the mechanism of interest. This contrasts with case-controlled studies that compare people with/without depression (regardless of morning activation); such designs could add mechanistic heterogeneity and divert signal from the process by which MADs relate to depression symptoms.

Aim 1 (observing mechanistic differences comparing ends of the MAD exposure spectrum): To characterize differences between dCGs who have MADs, compared with "morning type" dCGs, with regard to: (A) daily patterns rumination and mood symptoms; (B) resting-state connectivity; and (C) rumination cue-related activation.

Hypotheses: The group with MADs will have relatively (A) greater rumination and depression symptoms; and (B) greater resting amygdala-PCC connectivity; and (C) exaggerated limbic, DMN, and FPCN responses to rumination cues.

Additional model testing: Unique from concurrent correlations, MADs will predict later rumination and depression symptoms.

Aim 2 (modifying target): Among dCGs with MADs, test the effects of an active experimental probe targeting morning activity engagement (SAMM), compared with a contact-time matched control condition, on self-reported and actigraphy measured MADs.

Hypotheses: Relative to the control condition, the active probe will be associated with decreased self-reported MADs and increased actigraphy-measured morning activity.

Aim 3 (modifying mechanism via target): (A) Test effects of the active vs. control probes on EMA-measured rumination, resting-state connectivity, and brain network responses to rumination cues. (B) Evaluate if the probe's effects are explained by increases in morning activation.

Hypotheses: SAMM (vs. control) will be associated with reduced rumination and changes in the biomarker pattern listed in Aim 1.

Additional model testing: Experimental effects will be mediated by morning activation increases.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years or older.
* Provide at least 15 hours/week of unpaid care to a patient with a dementia diagnosis.
* Reporting stress or strain delivering care
* No or stable pharmacotherapy for depression
* Meets screening definition for having morning activation difficulty or a definite morning types per the Composite Morningness Questionnaire (CMQ)

Exclusion Criteria:

* Unsafe or unable to undergo MRI
* Active Cognitive Behavioral Therapy for mood or insomnia
* Probable dementia diagnosis
* Deadly illness or plans to leave the study area
* Current active substance use disorder

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in rumination at 6-months | Baseline, continuously up to weekly for 6-weeks, and follow-up (6 months)
  Rumination will be measured using the rumination subscale of the Behavioral Activation Scale for Depression (BASD). There is a minimum possible score of 0 and a maximum possible score of 24 with higher scores indicating higher [worse] rumination. This measure will be accessed via Ecological Momentary Assessment (EMA). A link will be sent to participant's mobile device by text message cuing participants to respond
Change from baseline in depressive symptoms at 6-months | Baseline, continuously up to weekly for 6-weeks, and follow-up (6 months)
  Depression will be measured using the Patient Health Questionnaire (PHQ-9). There is a minimum possible score of 0 and a maximum possible score of 27 with higher scores indicating higher [worse] depression.
Change from baseline in anxiety symptoms at 6-months | Baseline, continuously up to weekly for 6-weeks, and follow-up (6 months)
  Anxiety will be measured using the Generalized Anxiety Disorder 7-Item Scale (GAD-7). There is a minimum possible score of 0 and a maximum possible score of 21 with higher scores indicating higher [worse] anxiety.
Change in objective Morning Activation Deficits (MADs) over 1 week | Continuously for up to 1-week at baseline
  Morning activation deficits (MADs), a common component of depression measurable as actigraphy assessed morning inactivity.
Change in self-report Morning Activation Deficits (MADs) at 6-months | Baseline, continuously up to weekly for 6-weeks, and follow-up (6 months)
  Morning Activation Deficits (MADs) will be assessed using the Composite Morningness Questionnaire (CMQ). There is a minimum possible score of 13 and a maximum possible score of 55 with higher scores indicating a higher degree or morningness.
Change in resting-state connectivity at 6-weeks | Baseline and 6-weeks
  Resting connectivity of the amygdala and ventral posterior cingulate cortex (PCC) structures will be measured by brain imaging conducted with a 7 Tesla scanner
Change in neurological response to rumination cues at 6 weeks | Baseline and 6-weeks
  Rumination-related brain activation in the Limbic (amygdala), default mode network (DMN), ventral posterior cingulate cortex (PCC), and Frontal Parietal Control Network (FPCN) will be measured by brain imaging conducted with a 7 Tesla scanner.

SECONDARY OUTCOMES:
Change in self-report nocturnal mentation at 6-months | Baseline, continuously up to weekly for 6-weeks, and follow-up (6 months)
  Nocturnal mentation will be assessed using the nocturnal mentation subscale of Dream Recall Frequency Scale. There is a minimum possible score of 0 and a maximum possible score of 24 with higher scores [better] indicating less negative thoughts/feelings.
Change in self-report reward anticipation at 6-months | Baseline, continuously up to weekly for 6-weeks, and follow-up (6 months)
  Reward anticipation will be assessed using the a custom measure (e.g., "How much do you anticipate that your upcoming activities/things you do will be rewarding?"). There is a minimum possible score of 0 and a maximum possible score of 27 with higher scores indicating a higher degree of reward anticipation.
Change in self-report apathy at 6-months | Baseline, continuously up to weekly for 6-weeks, and follow-up (6 months)
  Apathy will be assessed using the Apathy Evaluation Scale. There is a minimum possible score of 18 and a maximum possible score of 72 with higher scores indicating a less apathy [better].
Change in morning light exposure at 6-weeks | Baseline and 6-weeks
  Light exposure will be assessed as lux levels in the morning from sensors on the actigraph
Change in cognitive functioning at 6-weeks | Baseline and 6-weeks
  Cognitive functioning will be measured by the Montreal Cognitive Assessment (MoCA), which was designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visual constructional skills, conceptual thinking, calculations, and orientation. There is a minimum possible score of 0 and maximum possible score of 30 with a higher score indicating better cognitive function. A score of 26 or above is considered normal.
Change in executive function at 6-weeks | Baseline and 6-weeks
  Executive function will be assessed by the Stroop Neuropsychological Screening Test, which was designed to measure inhibition. Participants have 120 seconds to name as many of the stimuli items as possible. Those with the ability to accurately employ inhibitory control, have better executive function. Scoring is based on percentiles and normative values, thus there is no minimum or maximum possible scores to report.
Change in cognitive functioning at 6-weeks | Baseline and 6-weeks
  Cognitive function will be assessed by the Trail-Making Test A and B, which was designed to measure executive function and memory. The Trail Making Test is scored by how long it takes to complete the test. The average time it takes to complete Part A is 29 seconds and a time greater than 78 seconds indicates impairment in these cognitive domains. The average time it takes to complete Part B is 75 seconds and a time greater than 273 seconds indicates impairment in these cognitive domains.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen F Smagula, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Western Behavioral Health, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No